CLINICAL TRIAL: NCT04772014
Title: The Addictive Potential of the E-Cigarette: Neurobiological, Sociological and Epidemiological Perspectives
Brief Title: Evaluation of the Addictive Potential of E-Cigarettes
Acronym: EVAPE
Status: Completed | Type: Observational
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Other Study IDs: EVAPE
Record Dates: First submitted 2020-12-30; First posted 2021-02-25 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Nicotine Use Disorder; Tobacco Use Disorder
Keywords: Nicotine; Electronic Nicotine Delivery Systems (ENDS); Addiction; Craving
MeSH Terms: conditions — Tobacco Use Disorder; Vaping; Behavior, Addictive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Salivary cotinine level
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- e-cigarette users: daily e-cigarette use (additional smoking of traditional tobacco cigarettes is not an exclusion criterion)
- nicotine-naïve: lifetime consumption of less than 20 cigarettes or e-cigarettes

SUMMARY:
This study will examine the subject matter from a neurobiological and a neuropsychological vantage point to ascertain whether the e-cigarette is potentially as addictive as the traditional tobacco cigarette.

DETAILED DESCRIPTION:
This project aims to examine the addictive potential of e-cigarettes through three different lenses, combining neurobiological, sociological and epidemiological research methods and levels of observation. The neurobiological perspective will investigate the rewarding effects of vaping, using neurobiological and neuropsychological measurements on e-cigarette users, as compared to nicotine-naïve participants.

The researchers will use established fMRI paradigms to measure the reward potential of e-cigarettes: First, craving will be investigated in an experimental approach by presenting conditioned stimuli to participants; and second, motivation for e-cigarettes compared to combustible cigarettes or money will be measured in an experimental work task. In addition, a dot-probe-task will be used in combination with eye-tracking to measure the attentional bias for e-cigarette stimuli. As part of the neuropsychological assessment outside the fMRI, the approach bias for smoking cues will also be investigated. The aim is to examine whether chronic use of e-cigarettes leads to similar conditioning processes and comparable aspects of motivation as that of traditional tobacco cigarettes.

The investigators will examine the punishment potential of e-cigarettes in a secondary research question, using questionnaires on withdrawal and on the consequences of smoking, both for traditional tobacco and for e-cigarettes.

The results of this project are relevant for the development of preventive healthcare and new treatment options. The neurobiological approach will also provide implications for individualized therapy by identifying consumer groups with different neuronal patterns.

ELIGIBILITY:
Inclusion Criteria:

* E-cigarette consumers: daily e-cigarette use (additional smoking of classic tobacco cigarettes is not an exclusion criterion)
* Nicotine Naïve: lifetime consumption of less than 20 cigarettes or e-cigarettes.
* normal or correctable eyesight
* sufficient ability to communicate with investigators and answer questions in both written and verbal format
* ability to provide fully informed consent and to use self-rating scales

Exclusion Criteria:

* common exclusion criteria for MRI (e.g. metal, claustrophobia, pregnancy)
* severe internal, neurological, and/or psychiatric comorbidities
* other Axis I mental disorders other than TUD or specific phobias within the last 12 months
* psychotropic medication within the last 14 days
* positive drug screening (opioids, benzodiazepines, barbiturates, cocaine, amphetamines)
* positive pregnancy test

The inclusion and exclusion criteria are checked in advance in a telephone screening. Smokers are asked not to smoke for eight hours before the examination.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: group 1: e-cigarette users, recruited from the local community group 2: nicotine-naïve (healthy controls), recruited from the local community
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Cue-reactivity [reward potency] | examination day 1 (single examination, no follow-up)
  fMRI to assess group differences in task-specific brain activation patterns using cue-reactivity task (Vollstädt-Klein et al. 2011)
Motivation [reward potency] | examination day 1 (single examination, no follow-up)
  fMRI to assess group differences in task-specific brain activation patterns using the MOTTA-task (Bühler et al. 2010);
Attentional-bias to smoking cues [reward potency] | examination day 1 (single examination, no follow-up)
  measured with reaction time differences (in milliseconds) using the smoke-related dot-probe task (Vollstadt-Klein et al. 2011) in combination with eye tracking and fMRI to assess group differences in task-specific eye movement and brain activation patterns
Approach-bias [reward potency] | examination day 1 (single examination, no follow-up)
  measured with reaction time differences (in milliseconds) using the smoking-related implicit association task (Wiers et al. 2016).
  [reaction time differences is not a change over time; it is measured during one experimental session]
Craving (CAS-CS) [reward potency] | examination day 1 (single examination, no follow-up)
  Assessment of self-reported craving for cigarette smoking using Craving Automatized Scale for Cigarette Smoking (CAS-CS): adapted from CAS-A (Vollstädt-Klein et al., 2015). 5 subscales (factors): Factor 1 ("only aware in hindsight") ranges from 0 to 35, factor 2 ("no deliberate decision") from 0 to 35, factor 3 ("contrary to intention") from 0 to 40, factor 4 ("no perception") from 0 to 20, and factor 5 ("no control") from 0 to 10, higher score means more habitual smoking.
Craving (QSU) [reward potency] | examination day 1
  Assessment of self-reported craving for cigarette smoking using Questionnaire of Smoking Urges (QSU, Müller et al. 2001); two subscales: "intention and desire to smoke / anticipation of pleasure from smoking" (range 11 - 77) and "anticipation of relief from negative affect and nicotine withdrawal / urgent and overwhelming desire to smoke" (range 10 - 70) high values represent high craving.
Craving (QSU) [reward potency] | examination day 2 (8-24 hours after examination day 1)
  Assessment of self-reported craving for cigarette smoking using Questionnaire of Smoking Urges (QSU, Müller et al. 2001); two subscales: "intention and desire to smoke / anticipation of pleasure from smoking" (range 11 - 77) and "anticipation of relief from negative affect and nicotine withdrawal / urgent and overwhelming desire to smoke" (range 10 - 70) high values represent high craving.
Craving (CAS-V) [reward potency] | examination day 1 (single examination, no follow-up)
  Assessment of self-reported craving for e-cigarettes using Craving Automatized Scale for Vaping (CAS-V): adapted from CAS-A (Vollstädt-Klein et al., 2015). 5 subscales (factors): Factor 1 ("only aware in hindsight") ranges from 0 to 35, factor 2 ("no deliberate decision") from 0 to 35, factor 3 ("contrary to intention") from 0 to 40, factor 4 ("no perception") from 0 to 20, and factor 5 ("no control") from 0 to 10, higher score means more habitual vaping.
Craving (QVC) [reward potency] | examination day 1
  Assessment of self-reported craving for e-cigarettes using Questionnaire of Vaping Craving (QVC; Dowd et al. 2018) 3 factors: Desire, Intention, Positive Outcome. Vaping craving ratings are made on a 7-point scale (1 = strongly disagree to 7 = strongly agree). high values represent high craving.
Craving (QVC) [reward potency] | examination day 2 (8-24 hours after examination day 1)
  Assessment of self-reported craving for e-cigarettes using Questionnaire of Vaping Craving (QVC; Dowd et al. 2018) 3 factors: Desire, Intention, Positive Outcome. Vaping craving ratings are made on a 7-point scale (1 = strongly disagree to 7 = strongly agree). high values represent high craving.

SECONDARY OUTCOMES:
Withdrawal symptoms [punishment potency] | examination day 1
  Assessment of Withdrawal symptoms of (e-cigarette) smoking using Wisconsin Smoking Withdrawal Scale (Welsch et al., 1999). 7 Subscales: anger, anxiety, concentration, craving, hunger, sadness, sleep. Each emotion is determined by the mean of each item that applies.
Withdrawal symptoms [punishment potency] | examination day 2 (8-24 hours after examination day 1)
  Assessment of Withdrawal symptoms of (e-cigarette) smoking using Wisconsin Smoking Withdrawal Scale (Welsch et al., 1999). 7 Subscales: anger, anxiety, concentration, craving, hunger, sadness, sleep. Each emotion is determined by the mean of each item that applies.
Negative consequences (SCQ) [punishment potency] | examination day 1 (single examination, no follow-up)
  Assessment of negative consequences of cigarette smoking using the Short Smoking Consequences Questionnaire (modified version of the SCQ (Brandon & Baker, 1991). Assesses cigarette smoking outcome expectancies among adolescents and young adults. 21-items, 10-point Likert scale (0=completely unlikely to 9=completely likely) to rate the likelihood of occurrence of each smoking consequence item. The four factors are consistent with the original SCQ subscales and include Negative Consequences (4 items), Positive Reinforcement (5 items), Negative Reinforcement (7 items), and Appetite-Weight Control (5 items). Higher scores stand for higher likelihood of consequences.
Negative consequences (VCQ) [punishment potency] | examination day 1 (single examination, no follow-up)
  Assessment of negative consequences of vaping e-cigarettes using the Short Vaping Consequences Questionnaire (modified version of the SCQ (Brandon & Baker, 1991). Assesses vaping e-cigarette outcome expectancies among adolescents and young adults. 21-items, 10-point Likert scale (0=completely unlikely to 9=completely likely) to rate the likelihood of occurrence of each vaping consequence item. The four factors are consistent with the original SCQ subscales and include Negative Consequences (4 items), Positive Reinforcement (5 items), Negative Reinforcement (7 items), and Appetite-Weight Control (5 items). Higher scores stand for higher likelihood of consequences.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Vollstädt-Klein, Principal Investigator — ZI Mannheim
Locations (1):
- Klinik für Abhängiges Verhalten, Zentralinstitut für Seelische Gesundheit, Mannheim, Germany

REFERENCES:
- [Derived] Vollstadt-Klein S, Grundinger N, Gorig T, Szafran D, Althaus A, Mons U, Schneider S. Study protocol: evaluation of the addictive potential of e-cigarettes (EVAPE): neurobiological, sociological, and epidemiological perspectives. BMC Psychol. 2021 Nov 18;9(1):181. doi: 10.1186/s40359-021-00682-8. PMID 34794514